CLINICAL TRIAL: NCT05932511
Title: Concentrated Ascorbic Acid in DMSO for Treatment of Squamous Cell Carcinoma of the Skin
Brief Title: Topical Ascorbic Acid for Treatment of Squamous Cell Skin Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Center for Biomedical Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCC_002
Record Dates: First submitted 2023-06-21; First posted 2023-07-06 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Squamous Cell Cancer; Squamous Cell Carcinoma; Skin Cancer; Non-melanoma Skin Cancer
Keywords: squamous cell cancer; skin cancer; non-melanoma skin cancer; squamous cell carcinoma
MeSH Terms: conditions — Neoplasms, Squamous Cell; Carcinoma, Squamous Cell; Skin Neoplasms | interventions — Ascorbic Acid; Dimethyl Sulfoxide

STUDY DESIGN:
Intervention Model Description: Open label pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 30% Ascorbic Acid in DMSO (Experimental): Topical application twice daily of 300ul 30% (w/v) solution of ascorbic acid in DMSO
  Interventions: Drug: 30% ascorbic acid in DMSO

INTERVENTIONS:
Drug: 30% ascorbic acid in DMSO — see above

SUMMARY:
Randomized comparative trial of a 30% solution of ascorbic acid in 95% dimethylsulfoxide applied topically twice a day for 8 weeks vs 5% imiquimod cream in the treatment of biopsy proven squamous cell carcinomas of the skin in otherwise healthy adult patients. Outcome measure was biopsy proven resolution of the carcinoma.

DETAILED DESCRIPTION:
Importance:

Skin cancer is the most common cancer in the United States, with more people diagnosed each year than all other cancers combined. Basal cell and squamous cell cancers are the most common forms with an estimated 6-7 million cases diagnosed annually. Costs of treating these cancers in the U.S. are estimated at $9-10 billion annually. Task force consensus guidelines suggest Mohs surgery as the treatment of choice, and as the single most precise and effective treatment method. However, cost and issues of cosmesis are principal disadvantages. Previous studies show the effectiveness of a topical solution of ascorbic acid in the treatment of BCC. This study extends previous work to evaluate efficacy in the treatment of SCC of the skin.

Objective:

To evaluate efficacy of a therapeutic regimen in treating squamous cell cancer, consisting of 30% ascorbic acid in 95% dimethylsulfoxide topically applied at home by patients twice a day for 8 weeks, vs 5% imiquimod cream which is an FDA approved treatment for SCC.

Design, Setting, and Participants:

This study was carried out in accordance with principles of the Declaration of Helsinki. Detailed informed consent was obtained from each patient.

Eligible participants of any age had histologically confirmed primary, previously untreated, nodular or superficial SCC. Patients with cancers larger than 2 cm or deeper than 2 mm were excluded from the study. Imiquimod was applied once daily for 5 days per week as per manufacturer instructions for treatment of SCC. Patients were randomly assigned to treatment group. Participants and outcome assessors were blinded to treatment protocol. Patients were seen at initial visit, 4 weeks, 8 weeks, and six weeks after treatment conclusion for final biopsy. The AA treatment was a solution while the IMQ a cream, however participants were simply told they would be receiving a topical treatment with instructions on how to apply, thus the blinding was intact.

Main Outcomes and Measures Number of lesions out that were cancer free after 8 wks of treatment.

ELIGIBILITY:
Inclusion Criteria: Presence of biopsy proven squamous cell cancer of the skin -

Exclusion Criteria: Previous history of malignancy, diabetes, immunocompromised

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Lesion Resolution | 8 weeks
  Number of lesions tumor free by 2 mm punch biopsy post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Biomedical Research,Inc., Boise, Idaho, United States